CLINICAL TRIAL: NCT04714320
Title: A Double-Blind, Placebo-Controlled, Phase 2 Study to Assess the Safety, Tolerability and Efficacy of IONIS-AGT-LRx, an Antisense Inhibitor of Angiotensinogen Production Administered Subcutaneously for 12 Weeks to Hypertensive Patients With Uncontrolled Blood Pressure
Brief Title: A Study to Assess the Safety, Tolerability and Efficacy of IONIS-AGT-LRx in Hypertensive Participants With Uncontrolled Blood Pressure
Acronym: ASTRAAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 757456-CS4
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: Hypertension; Hypertensive; AGT; Angiotensinogen; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pooled Placebo (Placebo Comparator): Participants received ISIS 757456 matching placebo subcutaneously once weekly for 12 weeks.
  Interventions: Drug: Placebo
- IONIS-AGT-LRx 80 mg (Experimental): Participants received ISIS 757456 80 milligrams (mg), subcutaneous (SC) injection, once weekly for 12 weeks.
  Interventions: Drug: IONIS-AGT-LRx
- IONIS-AGT-LRx 120 mg (Experimental): Participants received ISIS 757456 120 mg, SC injection, once weekly for 12 weeks.
  Interventions: Drug: IONIS-AGT-LRx

INTERVENTIONS:
Drug: Placebo — ISIS 757456 matching placebo administered by SC injection.
  Arms: Pooled Placebo
Drug: IONIS-AGT-LRx — IONIS-AGT-LRx administered by SC injection.
  Other Names: ISIS 757456
  Arms: IONIS-AGT-LRx 120 mg; IONIS-AGT-LRx 80 mg

SUMMARY:
The purpose of this study was to evaluate the effect of IONIS-AGT-LRx compared to placebo on seated automated office systolic blood pressure (SBP) from baseline to Study Day 85 in uncontrolled hypertensive participants on ≥ 3 antihypertensive medications and to evaluate the effect of IONIS-AGT-LRx on ambulatory blood pressure, seated automated office SBP, seated automated office diastolic blood pressure (DBP), and plasma angiotensinogen (AGT) at each scheduled visit in uncontrolled hypertensive participants on ≥ 3 antihypertensive medications.

DETAILED DESCRIPTION:
This was a phase 2, double-blind, randomized, placebo-controlled study in up to 160 participants. Participants were randomized in a 2:1 ratio and received a once-weekly subcutaneous (SC) treatment with either IONIS-AGT-LRx or matching placebo. The length of participation in the study was approximately 31 weeks, which included an up to 6-week screening period, a 12-week treatment period, and a 13-week post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18-80 inclusive and weighing ≥ 50 kilograms (kg) at the time of informed consent
* Females: must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal
* Males must be abstinent, surgically sterile or if engaged in sexual relations with a woman of childbearing potential (WOCBP), a highly effective contraceptive method must be used
* Body mass index (BMI) ≤ 45.0 kilograms per square meter (kg/m^2)
* At screening, the participant must have been on a stable, maximally tolerated regimen (per Investigator judgement) of 3 or more antihypertensive medications for at least 1 month prior to screening and will be required to maintain this regimen throughout the study. The combination of antihypertensive medications must be in the following categories: a) angiotensin-converting enzyme inhibitor (ACEi) or angiotensin II receptor blocker (ARB), b) beta blocker: c) calcium channel blocker d) diuretic, e) alpha-1 blocker f) centrally acting sympatholytic agent or g) direct acting vasodilators (e.g. hydralazine)

Exclusion Criteria:

* Clinically significant abnormalities in screening laboratory results, medical history according to Investigator judgment
* History of secondary hypertension (HTN) including, but not limited to any of the following: renovascular HTN (unilateral or bilateral renal artery stenosis), coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, and drug-induced HTN
* The use of the following at time of screening and during the course of the study:

  * Other medications for the treatment of HTN (e.g., minoxidil, diazoxide, renin inhibitors)
  * Medications that may cause hyperkalemia unless on a stable dose at least 1 month prior to the screening visit and no known history of hyperkalemia per Investigator judgement
  * Use of oral anticoagulants, unless stable for 4 weeks prior to the first dose of study drug and regular monitoring must be performed per clinical practice during the study unless the participant is receiving vitamin K agonists. If the participant is receiving vitamin K antagonists (e.g., warfarin) international normalized ratio (INR) should be in therapeutic range, as established by the Investigator, for 4 weeks prior to the first dose
  * Chronic administration of non-steroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase 2 (COX-2) inhibitors (except aspirin for cardiovascular disease provided the total daily dose does not exceed 325 mg)
* History of bleeding diathesis, coagulopathy, immune thrombocytopenic purpura (ITP), thrombotic cytopenic purpura (TTP), or any qualitative or quantitative platelet defect
* Unstable/underlying known cardiovascular disease defined as:

  * Any history of congestive heart failure (New York Heart Association [NYHA] Class III-IV)
  * Any history of previous myocardial infarction, coronary revascularization, unstable or stable angina pectoris ˂ 1 year prior to screening
  * Any hemodynamically unstable atrial or ventricular arrhythmias
  * Significant uncorrected valvular heart disease
  * Any history of stroke or transient ischemic attack < 1 year prior to screening
* A cardiac valve repair, cardiac device implantation, and/or a hospitalization for heart failure within 3 months of screening
* Participant works nighttime shifts (e.g., 11 PM to 7 AM)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (48):
  - Pinnacle Research Group, Anniston, Alabama
  - Central Research Associates, Inc., Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Cahaba Research, Inc., Pelham, Alabama
  - Syed Research Consultants LLC, Sheffield, Alabama
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - RESPIRE Research, La Mesa, California
  - Clinical Trials Research, Lincoln, California
  - Catalina Research Institute, Montclair, California
  - San Fernando Valley Health Institute, Van Nuys, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Chase Medical Research LLC, Waterbury, Connecticut
  - ALL Medical Research, LLC, Cooper City, Florida
  - Nature Coast Clinical Research - Crystal River, Crystal River, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Canvas Clinical Research, Lake Worth, Florida
  - Allied Biomedical Research Institute, Inc., Miami, Florida
  - AMPM Research Clinic, Miami Gardens, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Ocala Research Institute, Ocala, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Gwinnett Research Institute, Buford, Georgia
  - Sandhill Research, LLC, Decatur, Georgia
  - Georgia Institute for Clinical Research, Marietta, Georgia
  - Eagle Clinical Research, Chicago, Illinois
  - Clinical Investigation Specialists, Inc. - Wauconda, Wauconda, Illinois
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Louisiana Heart Center, Slidell, Louisiana
  - Clinical Trials of America, LLC - Monroe, LA, West Monroe, Louisiana
  - BioPharm Clinical Research, Caro, Michigan
  - Palm Research Center, Inc., Las Vegas, Nevada
  - NY Scientific, Brooklyn, New York
  - Summit Research Group, LLC, Stow, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Health Concepts Research, Rapid City, South Dakota
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - North Texas Research Associates, Allen, Texas
  - Juno Research, LL, Houston, Texas
  - Protenium Clinical Research, LLC, Hurst, Texas
  - Laguna Clinical Research Associates, Laredo, Texas
  - Kalo Clinical Research, Salt Lake City, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - TPMG Clinical Research, Williamsburg, Virginia
- Canada (2):
  - Ecogene-21, Chicoutimi, Quebec
  - CardioVasc HR, Saint-Jean-sur-Richelieu, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigative sites in the US and Canada from 28 April 2021 to 03 October 2022.
Pre-assignment Details: Participants with uncontrolled hypertension who were on ≥ 3 antihypertensive medications were enrolled and randomized to receive either ISIS 757456 80 mg, ISIS 757456 120 mg or ISIS 757456 matched placebo for a 12-week treatment period.
Groups:
- Pooled Placebo: Participants received ISIS 757456 matching placebo, subcutaneous (SC) injection, once weekly for 12 weeks.
- IONIS-AGT-LRx 80 mg: Participants received ISIS 757456 80mg, SC injection, once weekly for 12 weeks.
Period: Overall Study
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Started | 53 | 54 | 53
Per Protocol Set (PPS) (PPS included all Full Analysis Set (FAS) participants who received at least 10 of the 12 doses of study drug, did not alter antihypertensive medications during the treatment period and prior to Day 85, and have no significant protocol deviations that would be expected to affect efficacy assessment.) | 45 | 45 | 46
Completed | 48 | 50 | 47
Not Completed | 5 | 4 | 6
Not completed — Voluntary Withdrawal | 4 | 1 | 2
Not completed — Adverse Event or Serious Adverse Event (SAE) | 0 | 0 | 1
Not completed — Reason Not Specified | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Population: FAS included all randomized participants who received at least 1 injection of study drug (ISIS 757456 or placebo) and had at least 1 post-baseline efficacy measurements.
Groups:
- Pooled Placebo: Participants received ISIS 757456 matching placebo, SC injection, once weekly for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg | Total
Number analyzed (Participants) | 53 | 54 | 53 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.29) | 64.0 (7.47) | 61.3 (9.17) | 62.8 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 32 | 97
  Male | 20 | 22 | 21 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 15 | 14 | 49
  Not Hispanic or Latino | 33 | 39 | 39 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 35 | 30 | 29 | 94
  Race: Black | 16 | 20 | 21 | 57
  Race: Asian | 0 | 1 | 2 | 3
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Race: Other Race | 1 | 0 | 0 | 1
  Race: Multiple Races | 0 | 3 | 0 | 3
Seated Automated Office Systolic Blood Pressure (SBP)- PPS [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] — Population: PPS included all FAS participants who received at least 10 of the 12 doses of study drug, did not alter antihypertensive medications during the treatment period and prior to Day 85, and have no significant protocol deviations that would be expected to affect efficacy assessment.
  millimeters of mercury (mmHg)
    number analyzed (Participants) | 45 | 45 | 46 | 136
    (all) | 148.8 (12.51) | 143.3 (10.29) | 144.0 (11.35) | 145.3 (11.59)
Seated Automated Office Diastolic Blood Pressure (DBP)- PPS [Mean (Standard Deviation); unit: mmHg] — Population: PPS included all FAS participants who received at least 10 of the 12 doses of study drug, did not alter antihypertensive medications during the treatment period and prior to Day 85, and have no significant protocol deviations that would be expected to affect efficacy assessment.
  mmHg
    number analyzed (Participants) | 45 | 45 | 46 | 136
    (all) | 82.5 (8.50) | 80.6 (10.18) | 81.7 (10.48) | 81.6 (9.72)
Seated Automated Office Systolic Blood Pressure (SBP) -FAS [Mean (Standard Deviation); unit: mmHg] — Population: FAS included all randomized participants who received at least 1 injection of study drug (ISIS 757456 or placebo) and had at least 1 post-baseline efficacy measurements.
  mmHg | 147.6 (13.92) | 143.6 (10.04) | 144.1 (11.42) | 145.1 (11.95)
Seated Automated Office Diastolic Blood Pressure (DBP) -FAS [Mean (Standard Deviation); unit: mmHg] — Population: FAS included all randomized participants who received at least 1 injection of study drug (ISIS 757456 or placebo) and had at least 1 post-baseline efficacy measurements.
  mmHg | 82.1 (8.91) | 81.5 (10.20) | 82.8 (10.32) | 82.1 (9.78)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Seated Automated Office SBP to Day 85
Time Frame: Baseline to Day 85
Population: PPS included all FAS participants who received at least 10 of the 12 doses of study drug, did not alter antihypertensive medications during the treatment period and prior to Day 85, and had no significant protocol deviations that would have been expected to affect efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 45 | 45 | 46
mmHg | -9 [-14 to -3] | -13 [-18 to -8] | -9 [-14 to -4]
Statistical Analysis 1: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change From Baseline in Seated Automated Office SBP to Day 85; Test type: Superiority; p = 0.135, ANCOVA — The stratification factor (screening estimated glomerular filtration rate (eGFR) status [<60 vs. ≥60 mL/min/1.73 m^2]), treatment received, and baseline measure were included in the analysis of covariate (ANCOVA) model as independent variables
Statistical Analysis 2: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change From Baseline in Seated Automated Office SBP to Day 85; Test type: Superiority; p = 0.867, ANCOVA — The stratification factor (screening eGFR status [<60 vs. ≥60 mL/min/1.73 m2]), treatment received, and baseline measure were included in the ANCOVA model as independent variables

2. Secondary Outcome: Absolute Concentration of Plasma AGT at Each Scheduled, Post-Baseline Visit
Time Frame: Days 15, 29, 43, 57, 71, 85, 92, 106, 120, 148, and 169
Population: PPS included all FAS participants who received at least 10 of the 12 doses of study drug, did not alter antihypertensive medications during the Treatment Period and prior to Study Day 85, and have no significant protocol deviations that would be expected to affect efficacy assessment. 'Number analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 45 | 45 | 46
nmol/L
  At Day 15: number analyzed (Participants) | 45 | 44 | 46
  At Day 15 | 878.36 (239.895) | 575.68 (248.708) | 446.29 (189.521)
  At Day 29 | 836.74 (228.202) | 388.61 (193.723) | 293.27 (129.051)
  At Day 43: number analyzed (Participants) | 44 | 45 | 45
  At Day 43 | 837.24 (251.610) | 319.86 (180.741) | 239.02 (133.633)
  At Day 57: number analyzed (Participants) | 45 | 44 | 43
  At Day 57 | 848.45 (256.088) | 303.03 (168.530) | 293.12 (157.651)
  At Day 71: number analyzed (Participants) | 43 | 43 | 45
  At Day 71 | 790.50 (256.568) | 308.99 (174.893) | 308.86 (156.533)
  At Day 85: number analyzed (Participants) | 45 | 44 | 45
  At Day 85 | 793.77 (202.796) | 328.28 (199.364) | 321.71 (176.356)
  At Day 92: number analyzed (Participants) | 42 | 44 | 42
  At Day 92 | 748.11 (204.231) | 330.68 (176.868) | 317.93 (159.204)
  At Day 106: number analyzed (Participants) | 42 | 42 | 44
  At Day 106 | 756.89 (212.891) | 429.04 (175.316) | 443.95 (196.226)
  At Day 120: number analyzed (Participants) | 39 | 44 | 43
  At Day 120 | 746.63 (190.789) | 531.33 (203.681) | 562.27 (202.035)
  At Day 148: number analyzed (Participants) | 41 | 42 | 42
  At Day 148 | 753.35 (186.906) | 658.33 (248.413) | 662.13 (130.207)
  At Day 169: number analyzed (Participants) | 43 | 42 | 43
  At Day 169 | 797.92 (238.442) | 676.60 (236.881) | 700.48 (195.702)

3. Secondary Outcome: Change From Baseline in Plasma AGT to Each Scheduled, Post-Baseline Visit
Time Frame: Baseline, Days 15, 29, 43, 57, 71, 85, 92, 106, 120, 148, and 169
Population: PPS included all FAS participants who received at least 10 of the 12 doses of study drug, did not alter antihypertensive medications during the treatment period and prior to Day 85, and had no significant protocol deviations that would have been expected to affect efficacy assessment. 'Number analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 45 | 45 | 46
nmol/L
  Baseline | 833.42 (196.561) | 877.70 (290.487) | 836.60 (189.204)
  Change From Baseline at Day 15: number analyzed (Participants) | 45 | 44 | 46
  Change From Baseline at Day 15 | 44.94 (137.033) | -303.67 (187.426) | -390.31 (189.039)
  Change From Baseline at Day 29 | 3.31 (132.768) | -489.09 (260.294) | -543.33 (211.294)
  Change From Baseline at Day 43: number analyzed (Participants) | 44 | 45 | 45
  Change From Baseline at Day 43 | 8.15 (152.008) | -557.84 (267.373) | -544.34 (227.409)
  Change From Baseline at Day 57: number analyzed (Participants) | 45 | 44 | 43
  Change From Baseline at Day 57 | 15.03 (182.246) | -577.72 (282.528) | -542.84 (223.631)
  Change From Baseline at Day 71: number analyzed (Participants) | 43 | 43 | 45
  Change From Baseline at Day 71 | -47.31 (239.488) | -578.49 (276.950) | -522.65 (216.465)
  Change From Baseline at Day 85: number analyzed (Participants) | 45 | 44 | 45
  Change From Baseline at Day 85 | -39.65 (171.289) | -544.60 (314.195) | -517.42 (230.730)
  Change From Baseline at Day 92: number analyzed (Participants) | 42 | 44 | 42
  Change From Baseline at Day 92 | -73.33 (153.744) | -542.20 (281.935) | -523.31 (219.037)
  Change From Baseline at Day 106: number analyzed (Participants) | 42 | 42 | 44
  Change From Baseline at Day 106 | -57.84 (169.818) | -449.05 (288.731) | -395.60 (218.864)
  Change From Baseline at Day 120: number analyzed (Participants) | 39 | 44 | 43
  Change From Baseline at Day 120 | -64.61 (131.455) | -341.33 (259.403) | -282.34 (182.477)
  Change From Baseline at Day 148: number analyzed (Participants) | 41 | 42 | 42
  Change From Baseline at Day 148 | -62.29 (153.117) | -225.14 (233.595) | -165.06 (139.585)
  Change From Baseline at Day 169: number analyzed (Participants) | 43 | 42 | 43
  Change From Baseline at Day 169 | -18.31 (170.377) | -189.48 (260.868) | -129.72 (146.013)
Statistical Analysis 1: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change From Baseline at Day 15; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change From Baseline at Day 15; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 29; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 29; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 43; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 43; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 57; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 57; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 71; Test type: Superiority; p < 0.001, Van Elteren — The stratification factor (screening eGFR status [<60 vs. ≥60 mL/min/1.73 m2]) and treatment received were included in the Van Elteren model as independent variables
Statistical Analysis 10: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 71; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 11: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 85; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 12: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 85; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 13: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 92; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 92; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 106; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 16: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 106; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 17: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 120; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 120; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 148; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 20: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 148; Test type: Superiority; p = 0.002, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 21: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 169; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 22: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 169; Test type: Superiority; p = 0.002, Van Elteren — [p-value comment as in outcome 3, analysis 9]

4. Secondary Outcome: Percent Change From Baseline in Plasma AGT at Each Scheduled, Post-Baseline Visit
Time Frame: Baseline, Days 15, 29, 43, 57, 71, 85, 92, 106, 120, 148, and 169
Population: PPS included all FAS participants who received at least 10 of 12 doses of study drug did not alter antihypertensive medications during treatment period & prior to Day 85 have no significant protocol deviations that would be expected to affect efficacy assessment. 'Number analyzed' indicates number of participants with data available for analysis at specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 45 | 45 | 46
percent change
  Percent Change from Baseline at Day 15: number analyzed (Participants) | 45 | 44 | 46
  Percent Change from Baseline at Day 15 | 5.6 (16.8) | -34.3 (17.2) | -46.4 (18.8)
  Percent Change from Baseline at Day 29 | 0.5 (16.7) | -54.4 (18.3) | -63.6 (17.5)
  Percent Change from Baseline at Day 43: number analyzed (Participants) | 44 | 45 | 45
  Percent Change from Baseline at Day 43 | 0.3 (18.6) | -62.4 (16.5) | -63.2 (20.4)
  Percent Change from Baseline at Day 57: number analyzed (Participants) | 45 | 44 | 43
  Percent Change from Baseline at Day 57 | 1.6 (21.1) | -63.7 (17.9) | -64.0 (18.3)
  Percent Change from Baseline at Day 71: number analyzed (Participants) | 43 | 43 | 45
  Percent Change from Baseline at Day 71 | -4.8 (25.5) | -63.3 (19.4) | -62.0 (19.0)
  Percent Change from Baseline at Day 85: number analyzed (Participants) | 45 | 44 | 45
  Percent Change from Baseline at Day 85 | -3.3 (19.6) | -59.2 (27.4) | -60.7 (23.1)
  Percent Change from Baseline at Day 92: number analyzed (Participants) | 42 | 44 | 42
  Percent Change from Baseline at Day 92 | -8.3 (19.5) | -60.0 (18.7) | -61.4 (19.0)
  Percent Change from Baseline at Day 106: number analyzed (Participants) | 42 | 42 | 44
  Percent Change from Baseline at Day 106 | -6.3 (20.4) | -47.6 (22.8) | -46.4 (21.9)
  Percent Change from Baseline at Day 120: number analyzed (Participants) | 39 | 44 | 43
  Percent Change from Baseline at Day 120 | -7.3 (14.9) | -36.3 (20.6) | -33.2 (20.0)
  Percent Change from Baseline at Day 148: number analyzed (Participants) | 41 | 42 | 42
  Percent Change from Baseline at Day 148 | -6.1 (20.0) | -22.8 (25.4) | -18.4 (15.9)
  Percent Change from Baseline at Day 169: number analyzed (Participants) | 43 | 42 | 43
  Percent Change from Baseline at Day 169 | -2.0 (19.8) | -18.3 (29.6) | -15.2 (17.3)
Statistical Analysis 1: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 15; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 15; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day at 29; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day at 29; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 43; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 6: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 43; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 7: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 57; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 57; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 71; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 10: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 71; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 11: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 85; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 12: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 85; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 13: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 92; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 3, analysis 9]
Statistical Analysis 14: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 92; Test type: Superiority; p < 0.001, Van Elteren — The stratification factor (screening eGFR status (<60 vs ≥60 mL/min/1.73 m2)) and treatment received were included in the Van Elteren model as independent variables
Statistical Analysis 15: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 106; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 4, analysis 14]
Statistical Analysis 16: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 106; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 4, analysis 14]
Statistical Analysis 17: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 120; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 120; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 148; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 148; Test type: Superiority; p = 0.005, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Percent Change from Baseline at Day 169; Test type: Superiority; p < 0.001, Van Elteren — [p-value comment as in outcome 4, analysis 14]
Statistical Analysis 22: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Percent Change from Baseline at Day 169; Test type: Superiority; p = 0.002, Van Elteren — [p-value comment as in outcome 4, analysis 14]

5. Secondary Outcome: Change From Baseline to Study Day 85 in 24-hour Mean SBP and Diastolic Blood Pressure (DBP) Measured by Ambulatory Blood Pressure Monitoring (ABPM)
Time Frame: Baseline, Day 85
Population: PPS included all FAS participants who received at least 10 of the 12 doses of study drug, did not alter antihypertensive medications during the Treatment Period and prior to Study Day 85, and have no significant protocol deviations that would be expected to affect efficacy assessment. 'Overall number of participants analyzed' indicates the number of participants with data available for the analysis of this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 34 | 35 | 36
mmHg
  Change from Baseline in 24-hour Mean SBP at Day 85 | -1.362 [-5.696 to 2.973] | -5.675 [-9.631 to -1.718] | -0.862 [-5.035 to 3.311]
  Change from Baseline in 24-hour Mean DBP at Day 85 | -1.667 [-4.201 to 0.867] | -4.406 [-6.725 to -2.087] | -2.792 [-5.214 to -0.369]
Statistical Analysis 1: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline in 24-hour Mean SBP at Day 85; Test type: Superiority; p = 0.094, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline in 24-hour Mean SBP at Day 85; Test type: Superiority; p = 0.842, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change From Baseline in 24-hour Mean DBP at Day 85; Test type: Superiority; p = 0.066, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change From Baseline in 24-hour Mean DBP at Day 85; Test type: Superiority; p = 0.442, ANCOVA — [p-value comment as in outcome 1, analysis 2]

6. Secondary Outcome: Percentage of Participants Who Achieved Seated Automated Office SBP ≤ 140 mmHg, DBP ≤ 90 mmHg, and Both at Each Scheduled Post-Baseline Visit
Time Frame: Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 106, 120, 148, and 169
Population: PPS analysis set was used. Participants with SBP ≤ 140 mmHg at baseline were excluded from this analysis. 'Overall number of participants analyzed' indicates the number of participants with data available for the analysis of this outcome measure. 'Number analyzed' indicates number of participants with data available for analysis at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 32 | 26 | 25
percentage of participants
  Percentage of Participants With SBP ≤ 140 mmHg at Day 8 | 37.5 | 38.5 | 40.0
  Percentage of Participants With SBP ≤ 140 mmHg at Day 15 | 31.3 | 53.8 | 40.0
  Percentage of Participants With SBP ≤ 140 mmHg at Day 22 | 31.3 | 65.4 | 40.0
  Percentage of Participants With SBP ≤ 140 mmHg at Day 29 | 46.9 | 53.8 | 40.0
  Percentage of Participants With SBP ≤ 140 mmHg at Day 36: number analyzed (Participants) | 31 | 25 | 25
  Percentage of Participants With SBP ≤ 140 mmHg at Day 36 | 48.4 | 60.0 | 52.0
  Percentage of Participants With SBP ≤ 140 mmHg at Day 43: number analyzed (Participants) | 32 | 26 | 24
  Percentage of Participants With SBP ≤ 140 mmHg at Day 43 | 40.6 | 69.2 | 45.8
  Percentage of Participants With SBP ≤ 140 mmHg at Day 50: number analyzed (Participants) | 31 | 26 | 24
  Percentage of Participants With SBP ≤ 140 mmHg at Day 50 | 58.1 | 57.7 | 41.7
  Percentage of Participants With SBP ≤ 140 mmHg at Day 57: number analyzed (Participants) | 32 | 26 | 23
  Percentage of Participants With SBP ≤ 140 mmHg at Day 57 | 46.9 | 53.8 | 56.5
  Percentage of Participants With SBP ≤ 140 mmHg at Day 64: number analyzed (Participants) | 32 | 25 | 22
  Percentage of Participants With SBP ≤ 140 mmHg at Day 64 | 59.4 | 36.0 | 68.2
  Percentage of Participants With SBP ≤ 140 mmHg at Day 71: number analyzed (Participants) | 31 | 25 | 25
  Percentage of Participants With SBP ≤ 140 mmHg at Day 71 | 48.4 | 48.0 | 56.0
  Percentage of Participants With SBP ≤ 140 mmHg at Day 78: number analyzed (Participants) | 30 | 26 | 24
  Percentage of Participants With SBP ≤ 140 mmHg at Day 78 | 56.7 | 50.0 | 58.3
  Percentage of Participants With SBP ≤ 140 mmHg at Day 85: number analyzed (Participants) | 32 | 25 | 24
  Percentage of Participants With SBP ≤ 140 mmHg at Day 85 | 40.6 | 64.0 | 33.3
  Percentage of Participants With SBP ≤ 140 mmHg at Day 92: number analyzed (Participants) | 29 | 25 | 21
  Percentage of Participants With SBP ≤ 140 mmHg at Day 92 | 55.2 | 52.0 | 23.8
  Percentage of Participants With SBP ≤ 140 mmHg at Day 106: number analyzed (Participants) | 29 | 23 | 23
  Percentage of Participants With SBP ≤ 140 mmHg at Day 106 | 55.2 | 60.9 | 56.5
  Percentage of Participants With SBP ≤ 140 mmHg at Day 120: number analyzed (Participants) | 27 | 25 | 23
  Percentage of Participants With SBP ≤ 140 mmHg at Day 120 | 51.9 | 48.0 | 43.5
  Percentage of Participants With SBP ≤ 140 mmHg at Day 148: number analyzed (Participants) | 29 | 25 | 23
  Percentage of Participants With SBP ≤ 140 mmHg at Day 148 | 44.8 | 48.0 | 34.8
  Percentage of Participants With SBP ≤ 140 mmHg at Day 169: number analyzed (Participants) | 30 | 24 | 24
  Percentage of Participants With SBP ≤ 140 mmHg at Day 169 | 50.0 | 58.3 | 37.5
  Percentage of Participants With DBP ≤ 90 mmHg at Day 8 | 81.3 | 73.1 | 72.0
  Percentage of Participants With DBP ≤ 90 mmHg at Day 15 | 78.1 | 80.8 | 88.0
  Percentage of Participants With DBP ≤ 90 mmHg at Day 22 | 87.5 | 88.5 | 72.0
  Percentage of Participants With DBP ≤ 90 mmHg at Day 29 | 81.3 | 88.5 | 80.0
  Percentage of Participants With DBP ≤ 90 mmHg at Day 36: number analyzed (Participants) | 31 | 25 | 25
  Percentage of Participants With DBP ≤ 90 mmHg at Day 36 | 83.9 | 92.0 | 92.0
  Percentage of Participants With DBP ≤ 90 mmHg at Day 43: number analyzed (Participants) | 32 | 26 | 24
  Percentage of Participants With DBP ≤ 90 mmHg at Day 43 | 90.6 | 84.6 | 79.2
  Percentage of Participants With DBP ≤ 90 mmHg at Day 50: number analyzed (Participants) | 31 | 26 | 24
  Percentage of Participants With DBP ≤ 90 mmHg at Day 50 | 87.1 | 96.2 | 83.3
  Percentage of Participants With DBP ≤ 90 mmHg at Day 57: number analyzed (Participants) | 32 | 26 | 23
  Percentage of Participants With DBP ≤ 90 mmHg at Day 57 | 90.6 | 80.8 | 82.6
  Percentage of Participants With DBP ≤ 90 mmHg at Day 64: number analyzed (Participants) | 32 | 25 | 22
  Percentage of Participants With DBP ≤ 90 mmHg at Day 64 | 96.9 | 80.0 | 86.4
  Percentage of Participants With DBP ≤ 90 mmHg at Day 71: number analyzed (Participants) | 31 | 25 | 25
  Percentage of Participants With DBP ≤ 90 mmHg at Day 71 | 93.5 | 84.0 | 92.0
  Percentage of Participants With DBP ≤ 90 mmHg at Day 78: number analyzed (Participants) | 30 | 26 | 24
  Percentage of Participants With DBP ≤ 90 mmHg at Day 78 | 93.3 | 84.6 | 79.2
  Percentage of Participants With DBP ≤ 90 mmHg at Day 85: number analyzed (Participants) | 32 | 25 | 24
  Percentage of Participants With DBP ≤ 90 mmHg at Day 85 | 81.3 | 88.0 | 83.3
  Percentage of Participants With DBP ≤ 90 mmHg at Day 92: number analyzed (Participants) | 29 | 25 | 21
  Percentage of Participants With DBP ≤ 90 mmHg at Day 92 | 82.8 | 88.0 | 85.7
  Percentage of Participants With DBP ≤ 90 mmHg at Day 106: number analyzed (Participants) | 29 | 23 | 23
  Percentage of Participants With DBP ≤ 90 mmHg at Day 106 | 86.2 | 95.7 | 82.6
  Percentage of Participants With DBP ≤ 90 mmHg at Day 120: number analyzed (Participants) | 27 | 25 | 23
  Percentage of Participants With DBP ≤ 90 mmHg at Day 120 | 81.5 | 72.0 | 95.7
  Percentage of Participants With DBP ≤ 90 mmHg at Day 148: number analyzed (Participants) | 29 | 25 | 23
  Percentage of Participants With DBP ≤ 90 mmHg at Day 148 | 82.8 | 80.0 | 95.7
  Percentage of Participants With DBP ≤ 90 mmHg at Day 169: number analyzed (Participants) | 30 | 24 | 24
  Percentage of Participants With DBP ≤ 90 mmHg at Day 169 | 86.7 | 83.3 | 87.5
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 8 | 37.5 | 34.6 | 36.0
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 15 | 28.1 | 50.0 | 36.0
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 22 | 28.1 | 65.4 | 36.0
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 29 | 46.9 | 50.0 | 40.0
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 36: number analyzed (Participants) | 31 | 26 | 25
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 36 | 45.2 | 57.7 | 52.0
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 43: number analyzed (Participants) | 32 | 26 | 24
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 43 | 40.6 | 65.4 | 41.7
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 50: number analyzed (Participants) | 31 | 26 | 24
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 50 | 58.1 | 57.7 | 37.5
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 57: number analyzed (Participants) | 32 | 26 | 23
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 57 | 46.9 | 50.0 | 52.2
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 64: number analyzed (Participants) | 32 | 25 | 22
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 64 | 59.4 | 36.0 | 63.6
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 71: number analyzed (Participants) | 31 | 25 | 25
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 71 | 48.4 | 44.0 | 52.0
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 78: number analyzed (Participants) | 30 | 26 | 24
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 78 | 56.7 | 46.2 | 54.2
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 85: number analyzed (Participants) | 32 | 25 | 24
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 85 | 40.6 | 60.0 | 33.3
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 92: number analyzed (Participants) | 29 | 25 | 21
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 92 | 51.7 | 48.0 | 23.8
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 106: number analyzed (Participants) | 29 | 23 | 23
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 106 | 55.2 | 60.9 | 52.2
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 120: number analyzed (Participants) | 27 | 25 | 23
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 120 | 51.9 | 44.0 | 39.1
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 148: number analyzed (Participants) | 29 | 25 | 23
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 148 | 37.9 | 44.0 | 34.8
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 169: number analyzed (Participants) | 30 | 24 | 24
  Percentage of Participants With SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 169 | 50.0 | 54.2 | 37.5
Statistical Analysis 1: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 8; Test type: Superiority; p = 0.834, Regression, Logistic — Stratification factor (screening eGFR status (<60 vs ≤ 60 mL/min/1.73 m2)), treatment received and baseline measure were included in the Logistic Regression model, firth correction was applied if quasi-complete separation of data points was detected
Statistical Analysis 2: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 8; Test type: Superiority; p = 0.945, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 15; Test type: Superiority; p = 0.208, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 15; Test type: Superiority; p = 0.740, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 22; Test type: Superiority; p = 0.019, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 22; Test type: Superiority; p = 0.560, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 29; Test type: Superiority; p = 0.903, Regression, Logistic — Stratification factor (screening eGFR status (<60 vs ≤ 60 mL/min/1.73 m2)), treatment received and baseline measure are included in Logistic Regression model, firth correction will be applied if quasi-complete separation of data points is detected
Statistical Analysis 8: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 29; Test type: Superiority; p = 0.268, Regression, Logistic — [p-value comment as in outcome 6, analysis 7]
Statistical Analysis 9: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 36; Test type: Superiority; p = 0.702, Regression, Logistic — Stratification factor (screening eGFR status (<60 vs ≤ 60 mL/min/1.73 m2)), treatment received and baseline measure were included in Logistic Regression model, firth correction was applied if quasi-complete separation of data points was detected
Statistical Analysis 10: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 36; Test type: Superiority; p = 0.885, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 11: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 43; Test type: Superiority; p = 0.066, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 12: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 43; Test type: Superiority; p = 0.783, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 13: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 50; Test type: Superiority; p = 0.456, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 14: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 50; Test type: Superiority; p = 0.102, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 15: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 57; Test type: Superiority; p = 0.668, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 16: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 57; Test type: Superiority; p = 0.454, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 17: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 64; Test type: Superiority; p = 0.044, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 18: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 64; Test type: Superiority; p = 0.704, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 19: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 71; Test type: Superiority; p = 0.878, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 20: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 71; Test type: Superiority; p = 0.681, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 21: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 78; Test type: Superiority; p = 0.199, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 22: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 78; Test type: Superiority; p = 0.602, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 23: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 85; Test type: Superiority; p = 0.135, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 24: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 85; Test type: Superiority; p = 0.407, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 25: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 92; Test type: Superiority; p = 0.795, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 26: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 92; Test type: Superiority; p = 0.036, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 27: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 106; Test type: Superiority; p = 0.915, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 28: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 106; Test type: Superiority; p = 0.957, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 29: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 120; Test type: Superiority; p = 0.804, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 30: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 120; Test type: Superiority; p = 0.775, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 31: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 148; Test type: Superiority; p = 0.801, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 32: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 148; Test type: Superiority; p = 0.329, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 33: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 169; Test type: Superiority; p = 0.882, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 34: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg at Day 169; Test type: Superiority; p = 0.235, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 35: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 8; Test type: Superiority; p = 0.505, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 36: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 8; Test type: Superiority; p = 0.436, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 37: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 15; Test type: Superiority; p = 0.637, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 38: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 15; Test type: Superiority; p = 0.254, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 39: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 22; Test type: Superiority; p = 0.848, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 40: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 22; Test type: Superiority; p = 0.240, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 41: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 29; Test type: Superiority; p = 0.382, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 42: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 29; Test type: Superiority; p = 0.935, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 43: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 36; Test type: Superiority; p = 0.278, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 44: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 36; Test type: Superiority; p = 0.211, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 45: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 43; Test type: Superiority; p = 0.562, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 46: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 43; Test type: Superiority; p = 0.250, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 47: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 50; Test type: Superiority; p = 0.114, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 48: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 50; Test type: Superiority; p = 0.550, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 49: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 57; Test type: Superiority; p = 0.423, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 50: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 57; Test type: Superiority; p = 0.422, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 51: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 64; Test type: Superiority; p = 0.073, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 52: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 64; Test type: Superiority; p = 0.278, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 53: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 71; Test type: Superiority; p = 0.338, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 54: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 71; Test type: Superiority; p = 0.969, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 55: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 78; Test type: Superiority; p = 0.489, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 56: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 78; Test type: Superiority; p = 0.156, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 57: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 85; Test type: Superiority; p = 0.389, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 58: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 85; Test type: Superiority; p = 0.775, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 59: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 92; Test type: Superiority; p = 0.437, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 60: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 92; Test type: Superiority; p = 0.618, Regression, Logistic
Statistical Analysis 61: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 106; Test type: Superiority; p = 0.079, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 62: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 106; Test type: Superiority; p = 0.349, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 63: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 120; Test type: Superiority; p = 0.580, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 64: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 120; Test type: Superiority; p = 0.106, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 65: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 148; Test type: Superiority; p = 0.955, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 66: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 148; Test type: Superiority; p = 0.134, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 67: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 169; Test type: Superiority; p = 0.933, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 68: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 90 mmHg at Day 169; Test type: Superiority; p = 0.502, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 69: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 8; Test type: Superiority; p = 0.653, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 70: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 8; Test type: Superiority; p = 0.816, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 71: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 15; Test type: Superiority; p = 0.184, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 72: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 15; Test type: Superiority; p = 0.765, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 73: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 22; Test type: Superiority; p = 0.009, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 74: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 22; Test type: Superiority; p = 0.578, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 75: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 29; Test type: Superiority; p = 0.725, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 76: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 29; Test type: Superiority; p = 0.287, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 77: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 36; Test type: Superiority; p = 0.705, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 78: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 36; Test type: Superiority; p = 0.975, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 79: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 43; Test type: Superiority; p = 0.118, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 80: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 43; Test type: Superiority; p = 0.959, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 81: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 50; Test type: Superiority; p = 0.413, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 82: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 50; Test type: Superiority; p = 0.043, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 83: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 57; Test type: Superiority; p = 0.849, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 84: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 57; Test type: Superiority; p = 0.662, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 85: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 64; Test type: Superiority; p = 0.047, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 86: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 64; Test type: Superiority; p = 0.950, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 87: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 71; Test type: Superiority; p = 0.656, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 88: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 71; Test type: Superiority; p = 0.922, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 89: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 78; Test type: Superiority; p = 0.143, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 90: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 78; Test type: Superiority; p = 0.452, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 91: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 85; Test type: Superiority; p = 0.231, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 92: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 85; Test type: Superiority; p = 0.405, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 93: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 92; Test type: Superiority; p = 0.718, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 94: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 92; Test type: Superiority; p = 0.053, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 95: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 106; Test type: Superiority; p = 0.893, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 96: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 106; Test type: Superiority; p = 0.662, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 97: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 120; Test type: Superiority; p = 0.688, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 98: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 120; Test type: Superiority; p = 0.611, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 99: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 148; Test type: Superiority; p = 0.907, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 100: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 148; Test type: Superiority; p = 0.699, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 101: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 169; Test type: Superiority; p = 0.802, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 102: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 140 mmHg and DBP ≤ 90 mmHg at Day 169; Test type: Superiority; p = 0.206, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]

7. Secondary Outcome: Percentage of Participants Who Achieved Seated Automated SBP ≤ 130 mmHg, DBP ≤ 80 mmHg, and Both at Each Scheduled Post-Baseline Visit
Time Frame: Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 106, 120, 148, and 169
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- IONIS-AGT-LRx 120 mg: Participants received ISIS 757456 120 mg, SC injection, once-weekly for 12 weeks.
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 45 | 45 | 46
percentage of participants
  Percentage of Participants With SBP ≤ 130 mmHg at Day 8 | 20.0 | 37.8 | 30.4
  Percentage of Participants With SBP ≤ 130 mmHg at Day 15 | 20.0 | 35.6 | 26.1
  Percentage of Participants With SBP ≤ 130 mmHg at Day 22: number analyzed (Participants) | 44 | 45 | 46
  Percentage of Participants With SBP ≤ 130 mmHg at Day 22 | 27.3 | 31.1 | 34.8
  Percentage of Participants With SBP ≤ 130 mmHg at Day 29 | 28.9 | 44.4 | 43.5
  Percentage of Participants With SBP ≤ 130 mmHg at Day 36: number analyzed (Participants) | 44 | 44 | 45
  Percentage of Participants With SBP ≤ 130 mmHg at Day 36 | 36.4 | 43.2 | 48.9
  Percentage of Participants With SBP ≤ 130 mmHg at Day 43: number analyzed (Participants) | 45 | 45 | 45
  Percentage of Participants With SBP ≤ 130 mmHg at Day 43 | 28.9 | 46.7 | 44.4
  Percentage of Participants With SBP ≤ 130 mmHg at Day 50: number analyzed (Participants) | 44 | 45 | 45
  Percentage of Participants With SBP ≤ 130 mmHg at Day 50 | 27.3 | 44.4 | 40.0
  Percentage of Participants With SBP ≤ 130 mmHg at Day 57: number analyzed (Participants) | 45 | 44 | 43
  Percentage of Participants With SBP ≤ 130 mmHg at Day 57 | 24.4 | 43.2 | 39.5
  Percentage of Participants With SBP ≤ 130 mmHg at Day 64: number analyzed (Participants) | 45 | 44 | 43
  Percentage of Participants With SBP ≤ 130 mmHg at Day 64 | 40.0 | 31.8 | 34.9
  Percentage of Participants With SBP ≤ 130 mmHg at Day 71: number analyzed (Participants) | 43 | 43 | 45
  Percentage of Participants With SBP ≤ 130 mmHg at Day 71 | 30.2 | 44.2 | 40.0
  Percentage of Participants With SBP ≤ 130 mmHg at Day 78: number analyzed (Participants) | 43 | 43 | 45
  Percentage of Participants With SBP ≤ 130 mmHg at Day 78 | 41.9 | 44.2 | 37.8
  Percentage of Participants With SBP ≤ 130 mmHg at Day 85: number analyzed (Participants) | 45 | 44 | 45
  Percentage of Participants With SBP ≤ 130 mmHg at Day 85 | 26.7 | 50.0 | 37.8
  Percentage of Participants With SBP ≤ 130 mmHg at Day 92: number analyzed (Participants) | 42 | 44 | 42
  Percentage of Participants With SBP ≤ 130 mmHg at Day 92 | 40.5 | 34.1 | 33.3
  Percentage of Participants With SBP ≤ 130 mmHg at Day 106: number analyzed (Participants) | 42 | 42 | 44
  Percentage of Participants With SBP ≤ 130 mmHg at Day 106 | 35.7 | 52.4 | 40.9
  Percentage of Participants With SBP ≤ 130 mmHg at Day 120: number analyzed (Participants) | 39 | 44 | 43
  Percentage of Participants With SBP ≤ 130 mmHg at Day 120 | 28.2 | 34.1 | 30.2
  Percentage of Participants With SBP ≤ 130 mmHg at Day 148: number analyzed (Participants) | 41 | 42 | 43
  Percentage of Participants With SBP ≤ 130 mmHg at Day 148 | 31.7 | 33.3 | 27.9
  Percentage of Participants With SBP ≤ 130 mmHg at Day 169: number analyzed (Participants) | 43 | 42 | 43
  Percentage of Participants With SBP ≤ 130 mmHg at Day 169 | 30.2 | 42.9 | 34.9
  Percentage of Participants With DBP ≤ 80 mmHg at Day 8 | 53.3 | 64.4 | 60.9
  Percentage of Participants With DBP ≤ 80 mmHg at Day 15 | 48.9 | 66.7 | 56.5
  Percentage of Participants With DBP ≤ 80 mmHg at Day 22: number analyzed (Participants) | 44 | 45 | 46
  Percentage of Participants With DBP ≤ 80 mmHg at Day 22 | 59.1 | 64.4 | 58.7
  Percentage of Participants With DBP ≤ 80 mmHg at Day 29 | 60.0 | 68.9 | 65.2
  Percentage of Participants With DBP ≤ 80 mmHg at Day 36: number analyzed (Participants) | 44 | 44 | 45
  Percentage of Participants With DBP ≤ 80 mmHg at Day 36 | 56.8 | 75.0 | 55.6
  Percentage of Participants With DBP ≤ 80 mmHg at Day 43: number analyzed (Participants) | 45 | 45 | 45
  Percentage of Participants With DBP ≤ 80 mmHg at Day 43 | 57.8 | 71.1 | 60.0
  Percentage of Participants With DBP ≤ 80 mmHg at Day 50: number analyzed (Participants) | 44 | 45 | 45
  Percentage of Participants With DBP ≤ 80 mmHg at Day 50 | 63.6 | 66.7 | 53.3
  Percentage of Participants With DBP ≤ 80 mmHg at Day 57: number analyzed (Participants) | 45 | 44 | 43
  Percentage of Participants With DBP ≤ 80 mmHg at Day 57 | 66.7 | 68.2 | 65.1
  Percentage of Participants With DBP ≤ 80 mmHg at Day 64: number analyzed (Participants) | 45 | 44 | 43
  Percentage of Participants With DBP ≤ 80 mmHg at Day 64 | 60.0 | 68.2 | 62.8
  Percentage of Participants With DBP ≤ 80 mmHg at Day 71: number analyzed (Participants) | 43 | 43 | 45
  Percentage of Participants With DBP ≤ 80 mmHg at Day 71 | 58.1 | 58.1 | 62.2
  Percentage of Participants With DBP ≤ 80 mmHg at Day 78: number analyzed (Participants) | 43 | 43 | 45
  Percentage of Participants With DBP ≤ 80 mmHg at Day 78 | 67.4 | 69.8 | 66.7
  Percentage of Participants With DBP ≤ 80 mmHg at Day 85: number analyzed (Participants) | 45 | 44 | 45
  Percentage of Participants With DBP ≤ 80 mmHg at Day 85 | 60.0 | 75.0 | 66.7
  Percentage of Participants With DBP ≤ 80 mmHg at Day 92: number analyzed (Participants) | 42 | 44 | 42
  Percentage of Participants With DBP ≤ 80 mmHg at Day 92 | 66.7 | 70.5 | 64.3
  Percentage of Participants With DBP ≤ 80 mmHg at Day 106: number analyzed (Participants) | 42 | 42 | 44
  Percentage of Participants With DBP ≤ 80 mmHg at Day 106 | 61.9 | 66.7 | 59.1
  Percentage of Participants With DBP ≤ 80 mmHg at Day 120: number analyzed (Participants) | 39 | 44 | 43
  Percentage of Participants With DBP ≤ 80 mmHg at Day 120 | 64.1 | 63.6 | 60.5
  Percentage of Participants With DBP ≤ 80 mmHg at Day 148: number analyzed (Participants) | 41 | 42 | 43
  Percentage of Participants With DBP ≤ 80 mmHg at Day 148 | 53.7 | 61.9 | 60.5
  Percentage of Participants With DBP ≤ 80 mmHg at Day 169: number analyzed (Participants) | 43 | 42 | 43
  Percentage of Participants With DBP ≤ 80 mmHg at Day 169 | 55.8 | 66.7 | 48.8
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 8 | 17.8 | 33.3 | 26.1
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 15 | 20.0 | 33.3 | 17.4
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 22: number analyzed (Participants) | 44 | 45 | 46
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 22 | 27.3 | 24.4 | 30.4
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 29 | 24.4 | 40.0 | 34.8
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 36: number analyzed (Participants) | 44 | 45 | 45
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 36 | 27.3 | 37.8 | 35.6
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 43: number analyzed (Participants) | 45 | 45 | 45
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 43 | 24.4 | 37.8 | 35.6
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 50: number analyzed (Participants) | 44 | 45 | 45
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 50 | 25.0 | 37.8 | 28.9
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 57: number analyzed (Participants) | 45 | 44 | 43
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 57 | 22.2 | 40.9 | 30.2
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 64: number analyzed (Participants) | 45 | 44 | 43
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 64 | 33.3 | 25.0 | 25.6
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 71: number analyzed (Participants) | 43 | 43 | 45
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 71 | 30.2 | 34.9 | 31.1
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 78: number analyzed (Participants) | 43 | 43 | 45
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 78 | 37.2 | 37.2 | 37.8
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 85: number analyzed (Participants) | 45 | 44 | 45
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 85 | 26.7 | 40.9 | 31.1
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 92: number analyzed (Participants) | 42 | 44 | 42
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 92 | 38.1 | 27.3 | 28.6
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 106: number analyzed (Participants) | 42 | 42 | 44
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 106 | 31.0 | 40.5 | 29.5
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 120: number analyzed (Participants) | 39 | 44 | 43
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 120 | 25.6 | 31.8 | 23.3
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 148: number analyzed (Participants) | 41 | 42 | 43
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 148 | 26.8 | 31.0 | 23.3
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 169: number analyzed (Participants) | 43 | 42 | 43
  Percentage of Participants With SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 169 | 27.9 | 38.1 | 27.9
Statistical Analysis 1: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 8; Test type: Superiority; p = 0.280, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 2: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 8; Test type: Superiority; p = 0.648, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 3: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 15; Test type: Superiority; p = 0.416, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 4: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 15; Test type: Superiority; p = 0.900, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 5: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 22; Test type: Superiority; p = 0.627, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 6: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 22; Test type: Superiority; p = 0.921, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 7: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 29; Test type: Superiority; p = 0.464, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 8: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 29; Test type: Superiority; p = 0.458, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 9: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 36; Test type: Superiority; p = 0.779, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 10: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 36; Test type: Superiority; p = 0.629, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 11: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 43; Test type: Superiority; p = 0.242, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 12: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 43; Test type: Superiority; p = 0.290, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 13: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 50; Test type: Superiority; p = 0.349, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 14: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 50; Test type: Superiority; p = 0.532, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 15: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 57; Test type: Superiority; p = 0.205, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 16: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 57; Test type: Superiority; p = 0.368, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 17: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 64; Test type: Superiority; p = 0.084, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 18: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 64; Test type: Superiority; p = 0.179, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 19: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 71; Test type: Superiority; p = 0.584, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 20: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 71; Test type: Superiority; p = 0.762, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 21: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 78; Test type: Superiority; p = 0.675, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 22: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 78; Test type: Superiority; p = 0.166, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 23: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 85; Test type: Superiority; p = 0.090, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 24: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 85; Test type: Superiority; p = 0.488, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 25: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 92; Test type: Superiority; p = 0.218, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 26: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 92; Test type: Superiority; p = 0.232, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 27: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 106; Test type: Superiority; p = 0.421, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 28: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 106; Test type: Superiority; p = 0.815, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 29: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 120; Test type: Superiority; p = 0.711, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 30: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 120; Test type: Superiority; p = 0.514, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 31: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 148; Test type: Superiority; p = 0.479, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 32: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 148; Test type: Superiority; p = 0.292, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 33: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 169; Test type: Superiority; p = 0.528, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 34: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg at Day 169; Test type: Superiority; p = 0.946, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 35: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 8; Test type: Superiority; p = 0.552, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 36: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 8; Test type: Superiority; p = 0.598, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 37: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 15; Test type: Superiority; p = 0.184, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 38: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 15; Test type: Superiority; p = 0.614, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 39: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 22; Test type: Superiority; p = 0.933, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 40: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 22; Test type: Superiority; p = 0.803, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 41: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 29; Test type: Superiority; p = 0.686, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 42: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 29; Test type: Superiority; p = 0.752, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 43: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 36; Test type: Superiority; p = 0.106, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 44: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 36; Test type: Superiority; p = 0.779, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 45: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 43; Test type: Superiority; p = 0.323, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 46: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 43; Test type: Superiority; p = 0.991, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 47: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 50; Test type: Superiority; p = 0.973, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 48: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 50; Test type: Superiority; p = 0.230, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 49: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 57; Test type: Superiority; p = 0.792, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 50: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 57; Test type: Superiority; p = 0.744, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 51: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 64; Test type: Superiority — Stratification factor (screening eGFR status (<60 vs ≤ 60 mL/min/1.73 m2)), treatment received and baseline measure were included in Logistic Regression model, firth correction was applied if quasi-complete separation of data points was detected; p = 0.925, Regression, Logistic
Statistical Analysis 52: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 64; Test type: Superiority; p = 0.991, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 53: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 71; Test type: Superiority — [test comment as in outcome 7, analysis 51]; p = 0.530, Regression, Logistic
Statistical Analysis 54: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 71; Test type: Superiority; p = 0.849, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 55: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 78; Test type: Superiority; p = 0.953, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 56: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 78; Test type: Superiority; p = 0.884, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 57: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 85; Test type: Superiority; p = 0.230, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 58: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 85; Test type: Superiority; p = 0.589, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 59: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 92; Test type: Superiority; p = 0.919, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 60: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 92; Test type: Superiority; p = 0.753, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 61: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 106; Test type: Superiority; p = 0.747, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 62: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 106; Test type: Superiority; p = 0.764, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 63: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 120; Test type: Superiority; p = 0.527, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 64: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 120; Test type: Superiority; p = 0.639, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 65: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 148; Test type: Superiority; p = 0.744, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 66: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 148; Test type: Superiority; p = 0.539, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 67: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 169; Test type: Superiority; p = 0.417, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 68: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office DBP ≤ 80 mmHg at Day 169; Test type: Superiority; p = 0.466, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 69: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 8; Test type: Superiority; p = 0.380, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 70: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 8; Test type: Superiority; p = 0.730, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 71: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 15; Test type: Superiority; p = 0.595, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 72: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 15; Test type: Superiority; p = 0.279, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 73: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 22; Test type: Superiority; p = 0.196, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 74: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 22; Test type: Superiority; p = 0.728, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 75: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 29; Test type: Superiority; p = 0.453, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 76: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 29; Test type: Superiority; p = 0.681, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 77: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 36; Test type: Superiority; p = 0.863, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 78: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 36; Test type: Superiority; p = 0.837, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 79: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 43; Test type: Superiority; p = 0.504, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 80: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 43; Test type: Superiority; p = 0.531, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 81: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 50; Test type: Superiority; p = 0.600, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 82: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 50; Test type: Superiority; p = 0.830, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 83: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 57; Test type: Superiority; p = 0.209, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 84: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 57; Test type: Superiority; p = 0.809, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 85: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 64; Test type: Superiority; p = 0.045, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 86: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 64; Test type: Superiority; p = 0.104, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 87: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 71; Test type: Superiority; p = 0.690, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 88: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 71; Test type: Superiority; p = 0.590, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 89: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 78; Test type: Superiority; p = 0.538, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 90: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 78; Test type: Superiority; p = 0.407, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 91: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 85; Test type: Superiority; p = 0.398, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 92: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 85; Test type: Superiority; p = 0.930, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 93: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 92; Test type: Superiority; p = 0.111, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 94: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 92; Test type: Superiority; p = 0.196, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 95: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 106; Test type: Superiority; p = 0.816, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 96: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 106; Test type: Superiority; p = 0.473, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 97: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 120; Test type: Superiority; p = 0.615, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 98: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 120; Test type: Superiority; p = 0.214, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 99: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 148; Test type: Superiority; p = 0.575, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 100: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 148; Test type: Superiority; p = 0.276, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 101: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 169; Test type: Superiority; p = 0.573, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]
Statistical Analysis 102: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Seated Automated Office SBP ≤ 130 mmHg and DBP ≤ 80 mmHg at Day 169; Test type: Superiority; p = 0.706, Regression, Logistic — [p-value comment as in outcome 6, analysis 9]

8. Secondary Outcome: Change From Baseline in Seated Automated Office SBP to Each Scheduled, Post-Baseline Visit
Time Frame: Baseline, Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 106, 120, 148, and 169
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 45 | 45 | 46
mmHg
  Change from Baseline at Day 8 | -7.98 (13.973) | -5.87 (12.427) | -4.78 (13.306)
  Change from Baseline at Day 15 | -7.38 (14.967) | -7.73 (13.768) | -4.11 (11.443)
  Change from Baseline at Day 22: number analyzed (Participants) | 44 | 45 | 46
  Change from Baseline at Day 22 | -9.50 (15.725) | -7.84 (16.100) | -6.80 (13.881)
  Change from Baseline at Day 29 | -9.49 (16.385) | -9.13 (14.258) | -6.91 (12.096)
  Change from Baseline at Day 36: number analyzed (Participants) | 44 | 44 | 45
  Change from Baseline at Day 36 | -11.48 (15.953) | -11.57 (13.971) | -6.40 (14.318)
  Change from Baseline at Day 43: number analyzed (Participants) | 45 | 45 | 45
  Change from Baseline at Day 43 | -9.31 (11.853) | -11.73 (15.193) | -7.24 (16.563)
  Change from Baseline at Day 50: number analyzed (Participants) | 44 | 45 | 45
  Change from Baseline at Day 50 | -10.93 (12.250) | -9.64 (17.112) | -6.13 (16.453)
  Change from Baseline at Day 57: number analyzed (Participants) | 45 | 44 | 43
  Change from Baseline at Day 57 | -10.13 (13.844) | -9.89 (14.257) | -7.47 (18.194)
  Change from Baseline at Day 64: number analyzed (Participants) | 45 | 44 | 43
  Change from Baseline at Day 64 | -13.31 (13.019) | -7.70 (14.305) | -8.19 (15.241)
  Change from Baseline at Day 71: number analyzed (Participants) | 43 | 43 | 45
  Change from Baseline at Day 71 | -12.26 (14.671) | -8.35 (15.426) | -5.71 (16.045)
  Change from Baseline at Day 78: number analyzed (Participants) | 43 | 43 | 45
  Change from Baseline at Day 78 | -14.19 (11.827) | -9.37 (16.435) | -8.22 (14.734)
  Change from Baseline at Day 85: number analyzed (Participants) | 45 | 44 | 45
  Change from Baseline at Day 85 | -9.64 (16.346) | -10.93 (15.319) | -6.98 (15.995)
  Change from Baseline at Day 92: number analyzed (Participants) | 42 | 44 | 42
  Change from Baseline at Day 92 | -11.76 (18.127) | -7.57 (15.855) | -6.57 (13.110)
  Change from Baseline at Day 106: number analyzed (Participants) | 42 | 42 | 44
  Change from Baseline at Day 106 | -12.14 (13.258) | -8.57 (16.476) | -6.61 (16.158)
  Change from Baseline at Day 120: number analyzed (Participants) | 39 | 44 | 43
  Change from Baseline at Day 120 | -9.36 (13.240) | -5.14 (15.514) | -5.14 (15.020)
  Change from Baseline at Day 148: number analyzed (Participants) | 41 | 42 | 43
  Change from Baseline at Day 148 | -9.07 (13.650) | -6.76 (15.637) | -4.30 (14.393)
  Change from Baseline at Day 169: number analyzed (Participants) | 43 | 42 | 43
  Change from Baseline at Day 169 | -9.23 (13.336) | -8.76 (16.798) | -2.02 (17.468)
Statistical Analysis 1: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 8; Test type: Superiority; p = 0.853, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 8; Test type: Superiority; p = 0.542, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.430, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.587, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 22; Test type: Superiority; p = 0.910, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 22; Test type: Superiority; p = 0.846, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 29; Test type: Superiority; p = 0.634, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 29; Test type: Superiority; p = 0.767, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 36; Test type: Superiority; p = 0.399, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 36; Test type: Superiority; p = 0.323, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 43; Test type: Superiority; p = 0.115, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 43; Test type: Superiority; p = 0.982, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 50; Test type: Superiority; p = 0.859, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 50; Test type: Superiority; p = 0.344, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 57; Test type: Superiority; p = 0.633, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 57; Test type: Superiority; p = 0.889, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 64; Test type: Superiority; p = 0.241, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 64; Test type: Superiority; p = 0.367, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 71; Test type: Superiority; p = 0.716, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 71; Test type: Superiority; p = 0.210, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 78; Test type: Superiority; p = 0.363, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 78; Test type: Superiority; p = 0.193, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 85; Test type: Superiority; p = 0.135, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 85; Test type: Superiority; p = 0.867, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 25: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 92; Test type: Superiority; p = 0.761, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 26: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 92; Test type: Superiority; p = 0.618, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 27: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 106; Test type: Superiority; p = 0.363, Van Elteren — The stratification factor (screening eGFR status (<60 vs ≥60 mL/min/1.73 m2)) and treatment received are included in the Van Elteren model as independent variables
Statistical Analysis 28: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 106; Test type: Superiority; p = 0.125, Van Elteren — [p-value comment as in outcome 8, analysis 27]
Statistical Analysis 29: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 120; Test type: Superiority; p = 0.435, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 30: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 120; Test type: Superiority; p = 0.413, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 31: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 148; Test type: Superiority; p = 0.658, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 32: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 148; Test type: Superiority; p = 0.275, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 33: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 169; Test type: Superiority; p = 0.578, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 34: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 169; Test type: Superiority; p = 0.114, ANCOVA — [p-value comment as in outcome 1, analysis 2]

9. Secondary Outcome: Change From Baseline in Seated Automated Office DBP to Each Scheduled, Post-Baseline Visit
Time Frame: Baseline, Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 106, 120, 148, and 169
Population: PPS included all FAS participants who received at least 10 of 12 doses of study drug, did not alter antihypertensive medications during treatment period and prior to Day 85,and had no significant protocol deviations that would have been expected to affect efficacy assessment. 'Number analyzed' is the number of participants with data available for analysis at the specified timepoint
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
Number analyzed (Participants) | 45 | 45 | 46
mmHg
  Change from Baseline at Day 8 | -5.07 [-8.20 to 1.94] | -3.47 [-6.44 to -0.49] | -4.25 [-7.31 to -1.19]
  Change from Baseline at Day 15 | -4.78 [-7.84 to -1.73] | -4.70 [-7.59 to -1.80] | -4.38 [-7.36 to -1.40]
  Change from Baseline at Day 22: number analyzed (Participants) | 44 | 45 | 46
  Change from Baseline at Day 22 | -6.05 [-9.48 to -2.62] | -5.62 [-8.78 to -2.45] | -4.31 [-7.57 to -1.04]
  Change from Baseline at Day 29 | -5.93 [-9.02 to -2.85] | -6.72 [-9.65 to -3.79] | -4.84 [-7.86 to -1.83]
  Change from Baseline at Day 36: number analyzed (Participants) | 44 | 44 | 45
  Change from Baseline at Day 36 | -4.87 [-8.03 to -1.72] | -6.32 [-9.32 to -3.33] | -3.90 [-6.98 to -0.82]
  Change from Baseline at Day 43: number analyzed (Participants) | 45 | 45 | 45
  Change from Baseline at Day 43 | -6.37 [-9.52 to -3.23] | -6.87 [-9.86 to -3.89] | -5.42 [-8.50 to -2.33]
  Change from Baseline at Day 50: number analyzed (Participants) | 44 | 45 | 45
  Change from Baseline at Day 50 | -4.72 [-7.64 to -1.81] | -5.99 [-8.74 to -3.24] | -3.29 [-6.13 to -0.45]
  Change from Baseline at Day 57: number analyzed (Participants) | 45 | 44 | 43
  Change from Baseline at Day 57 | -8.06 [-11.14 to -4.97] | -7.90 [-10.84 to -4.97] | -6.26 [-9.38 to -3.14]
  Change from Baseline at Day 64: number analyzed (Participants) | 45 | 44 | 43
  Change from Baseline at Day 64 | -7.52 [-10.31 to -4.72] | -5.73 [-8.40 to -3.06] | -5.26 [-8.03 to -2.48]
  Change from Baseline at Day 71: number analyzed (Participants) | 43 | 43 | 45
  Change from Baseline at Day 71 | -7.59 [-10.54 to -4.64] | -5.36 [-8.16 to -2.56] | -6.46 [-9.32 to -3.59]
  Change from Baseline at Day 78: number analyzed (Participants) | 43 | 43 | 45
  Change from Baseline at Day 78 | -7.83 [-10.79 to -4.87] | -6.11 [-8.91 to -3.31] | -5.87 [-8.74 to -2.99]
  Change from Baseline at Day 85: number analyzed (Participants) | 45 | 44 | 45
  Change from Baseline at Day 85 | -5.20 [-8.24 to -2.16] | -6.78 [-9.68 to -3.88] | -6.13 [-9.11 to -3.14]
  Change from Baseline at Day 92: number analyzed (Participants) | 42 | 44 | 42
  Change from Baseline at Day 92 | -6.13 [-9.37 to -2.90] | -5.82 [-8.85 to -2.79] | -4.87 [-8.11 to -1.62]
  Change from Baseline at Day 106: number analyzed (Participants) | 42 | 42 | 44
  Change from Baseline at Day 106 | -5.61 [-8.95 to -2.27] | -5.94 [-9.08 to -2.79] | -4.85 [-8.01 to -1.68]
  Change from Baseline at Day 120: number analyzed (Participants) | 39 | 44 | 43
  Change from Baseline at Day 120 | -5.50 [-8.77 to -2.24] | -3.50 [-6.36 to -0.63] | -4.68 [-7.67 to -1.70]
  Change from Baseline at Day 148: number analyzed (Participants) | 41 | 42 | 43
  Change from Baseline at Day 148 | -4.67 [-8.18 to -1.71] | -4.80 [-7.93 to -1.67] | -3.86 [-7.17 to -0.55]
  Change from Baseline at Day 169: number analyzed (Participants) | 43 | 42 | 43
  Change from Baseline at Day 169 | -4.07 [-7.39 to -0.75] | -5.34 [-8.43 to -2.26] | -1.54 [-4.79 to 1.72]
Statistical Analysis 1: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 8; Test type: Superiority; p = 0.378, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 8; Test type: Superiority; p = 0.648, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.961, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.817, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 22; Test type: Superiority; p = 0.823, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 22; Test type: Superiority; p = 0.362, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 29; Test type: Superiority; p = 0.660, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 29; Test type: Superiority; p = 0.539, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 36; Test type: Superiority; p = 0.430, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 36; Test type: Superiority; p = 0.594, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 43; Test type: Superiority; p = 0.783, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 43; Test type: Superiority; p = 0.599, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 50; Test type: Superiority; p = 0.454, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 50; Test type: Superiority; p = 0.394, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 57; Test type: Superiority; p = 0.930, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 57; Test type: Superiority; p = 0.313, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 64; Test type: Superiority; p = 0.276, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 64; Test type: Superiority; p = 0.168, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 71; Test type: Superiority; p = 0.199, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 71; Test type: Superiority; p = 0.506, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 78; Test type: Superiority; p = 0.320, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 78; Test type: Superiority; p = 0.250, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 85; Test type: Superiority; p = 0.373, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 85; Test type: Superiority; p = 0.597, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 25: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 92; Test type: Superiority; p = 0.867, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 26: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 92; Test type: Superiority; p = 0.500, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 27: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 106; Test type: Superiority; p = 0.863, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 28: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 106; Test type: Superiority; p = 0.681, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 29: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 120; Test type: Superiority; p = 0.262, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 30: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 120; Test type: Superiority; p = 0.645, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 31: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 148; Test type: Superiority; p = 0.947, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 32: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 148; Test type: Superiority; p = 0.665, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 33: Comparison: Pooled Placebo vs IONIS-AGT-LRx 80 mg; Change from Baseline at Day 169; Test type: Superiority; p = 0.498, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 34: Comparison: Pooled Placebo vs IONIS-AGT-LRx 120 mg; Change from Baseline at Day 169; Test type: Superiority; p = 0.173, ANCOVA — [p-value comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to end of post-treatment period (up to 25 weeks)
Description: Safety set included all randomized participants that received at least 1 dose of study drug.
Arm/Group | Pooled Placebo | IONIS-AGT-LRx 80 mg | IONIS-AGT-LRx 120 mg
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/54 | 1/53
Serious Adverse Events (participants affected / at risk) | 1/53 | 2/54 | 1/53
Other Adverse Events (participants affected / at risk) | 9/53 | 18/54 | 14/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=53) | IONIS-AGT-LRx 80 mg (N=54) | IONIS-AGT-LRx 120 mg (N=53)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=53) | IONIS-AGT-LRx 80 mg (N=54) | IONIS-AGT-LRx 120 mg (N=53)
Nausea (Gastrointestinal disorders) | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2
Injection site erythema (General disorders) | 0 | 2 | 3
COVID-19 (Infections and infestations) | 1 | 2 | 3
Urinary tract infection (Infections and infestations) | 2 | 5 | 3
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Headache (Nervous system disorders) | 4 | 1 | 2
Hypertension (Vascular disorders) | 3 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT04714320/Prot_SAP_001.pdf